CLINICAL TRIAL: NCT00255086
Title: The Effect of Memantine on Brain Structure and Chemistry in Alzheimer's Disease Patients: A Randomized, Placebo-Controlled, 52-Week Clinical Trial
Brief Title: The Effect of Memantine on Brain Structure and Chemistry in Alzheimer's Disease Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Palo Alto Veterans Institute for Research (Other); Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Jerome A Yesavage,, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 95722
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-02

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Memantine (Experimental): 10mg Memantine
  Interventions: Drug: Memantine
- Control (Placebo Comparator): 10 mg Placebo pill
  Interventions: Drug: Placebo pill

INTERVENTIONS:
Drug: Memantine — 10mg Memantine
  Other Names: Namenda
  Arms: Memantine
Drug: Placebo pill — 10mg placebo pill
  Other Names: placebo
  Arms: Control

SUMMARY:
The aim of the proposed study is to determine if the NMDA receptor antagonist memantine has a neuroprotective effect on magnetic resonance spectroscopic imaging (MRS) measures of brain NAA and magnetic resonance imaging (MRI) volumetric measures of hippocampal volume. In secondary analyses, we will determine if measures of clinical stabilization produced by memantine in the treatment of Alzheimer's disease (AD) parallels stabilization of MRS measures of brain NAA and MRI volumetric measures of hippocampal volume.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is the most common form of dementia. Currently, there are more than 4 million individuals with dementia in the United States with at least 400,000 deaths annually. AD is a progressive, neurodegenerative disorder, characterized neuropathologically by widespread neuronal loss, presence of neurofibrillary tangles, and deposits of beta amyloid in cerebral blood vessels and neuritic plaques. Since the medial-temporal lobes, hippocampus, and association cortex are significantly impacted it is not surprising that the primary symptom of AD is a decline in cognitive functioning that leads to marked impairment in daily functioning. In particular, memory impairments, visuospatial decline, language difficulties, and loss of executive function are central cognitive symptoms of this illness. Behavioral disturbances such as agitation and hallucinations often accompany disease progression. The illness lasts approximately 7 to 10 years, with patients requiring total care in the latter stages. Thus, AD places a tremendous emotional and economic burden on both patients and their caregivers. Beyond a cure, therapeutic approaches which would alleviate the symptoms or delay progression could be of substantial psychological and economic benefit. Recent placebo controlled clinical trials have shown memantine to be efficacious in the treatment of patients with moderate to severe AD.

The aim of the proposed study is to determine if the NMDA receptor antagonist memantine has a neuroprotective effect on magnetic resonance spectroscopic imaging (MRS) measures of brain NAA and magnetic resonance imaging (MRI) volumetric measures of hippocampal volume. In secondary analyses, we will determine if measures of clinical stabilization produced by memantine in the treatment of Alzheimer's disease (AD) parallels stabilization of MRS measures of brain NAA and MRI volumetric measures of hippocampal volume.

ELIGIBILITY:
Inclusion Criteria:1. Dementia criteria by DSM-IV.

2. 50-95 years of age inclusive.

3. MMSE at screen and baseline 7-28 inclusive.

4. Conversant in English.

5. Caregiver/study partner willing to participate, supervise the patient and be available for administration of study medication.

6. Able to ingest oral medication. Exclusion Criteria:1. History of clinically significant stroke without substantial recovery.

2. Neurological or medical conditions causing significant disability independent of dementia.

3. Parkinson's disease.

4. History in past two years of focal brain lesion, head injury with loss of consciousness or DSM-IV criteria for any major psychiatric disorder including psychosis, major depression, bipolar disorder, alcohol or substance abuse.

5. Dementia due to Korsakoff's syndrome or infectious diseases such as Creutzfeldt-Jakob disease, herpes, encephalitis, or human immunodeficiency virus.

6. Sensory impairment that would prevent subject from participating in or cooperating with the protocol.

7. Significant clinical disorder or laboratory finding that renders the subject unsuitable for receiving an investigational drug including: clinically significant or unstable hematologic, hepatic, cardiovascular, pulmonary, gastrointestinal, endocrine, metabolic, renal, or other systemic disease or laboratory abnormality.

8. Clinical contraindication to the use of memantine (e.g., hypersensitivity).

9. History of seizure within past 5 years prior to screening.

10. Platelet count < 100,000/mm3.

11. History of claustrophobia

12. Presence of metallic implants such as pacemakers, surgical aneurysm clips, or known metal fragments embedded in the body

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-05; Primary Completion 2009-06 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Wesson Ashford Jr., MD, PhD, Study Director — Stanford University; Jerome A Yesavage, Principal Investigator — Stanford University
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 17 subjects were randomized. All subjects had completed all participation by October, 2008. All were recruited at VA Palo Alto Health Care System.
Groups:
- Memantine: 10mg Memantine
  Memantine
- Control: Participants were given Placebo
Period: Overall Study
Arm/Group | Memantine | Control
Started | 9 | 8
Completed | 7 | 6
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Population: Per protocol, only participants who completed the study were evaluable for baseline characteristics.
Groups:
- Control: 10mg Placebo pill
- Total: Total of all reporting groups
Arm/Group | Memantine | Control | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Full Range); unit: years] | 76.5 [50 to 90] | 75.4 [50 to 90] | 75.9 [50 to 90]
Sex/Gender, Customized [Number; unit: participants]
  Female | 1 | 4 | 5
  Male | 6 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: NAA/Cr Ratio
Description: To determine if memantine has a neuroprotective effect on magnetic resonance spectroscopic imaging (MRS) measures of hippocampal n-acetyl aspartate (NAA) and magnetic resonance imaging volumetric measures (MRI) of hippocampal volume.
Time Frame: Baseline; Year 1
Population: Participants who could tolerate study medication and who completed the study were included in the analysis.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Memantine | Control
Number analyzed (Participants) | 4 | 6
Ratio
  Baseline | 1.47 (0.11) | 1.38 (0.10)
  Year 1 | 1.62 (0.14) | 1.41 (0.10)

2. Secondary Outcome: Mean Change on the ADAS-Cog Score After 1 Year
Description: Progression of cognitive functioning as measured by performance on the Alzheimer's Disease (AD) Assessment Scale-cognitive subscale (ADAS-Cog). ADAS-cog is the most popular cognitive testing instrument used in clinical trials of nootropics, and measures disturbances of of memory, language, praxis, attention and other cognitive abilities which are often referred to as the core symptoms of AD. Responses are summed for an overall score which can range from 0-70. The greater the dysfunction, the higher the score. A typical score for a person without dementia is 5.
Time Frame: Baseline; Year 1
Population: Participants who could tolerate study medication and who completed the study were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine | Control
Number analyzed (Participants) | 4 | 6
units on a scale
  Baseline | 44.67 (10.30) | 49.17 (8.37)
  1 Year | 45.75 (7.99) | 50.39 (8.88)

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- Control: Participants were given matching placebo
Arm/Group | Memantine | Control
Serious Adverse Events (participants affected / at risk) | 1/9 | 2/8
Other Adverse Events (participants affected / at risk) | 4/9 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (N=9) | Control (N=8)
Cardiac Arrythmia (Cardiac disorders) | 1 (1) | 0 (0) — Not related to study medication; incident occurred before medication was started; family notified researcher of problem and subject withdrawn.
Crohn's disease flare-ups (Gastrointestinal disorders) | 0 (0) | 1 (1) — Not related to study medication (subject was on placebo). Notified by patient. Hospitalized, treated and released, continued with study.
complications due to type II diabetes (Endocrine disorders) | 0 (0) | 1 (1) — Not related to study medication (on placebo). Hospitalized, withdrawn from study. Later died.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (N=9) | Control (N=8)
Tattoo eyeliner (Eye disorders) | 1 (1) | 0 (0) — Study requirement is MRI. Unable to complete study procedures due to tattoo eyeliner so subject was withdrawn by the PI. Not study related.
Lethargy (Psychiatric disorders) | 1 (1) | 0 (0) — Subject discontinued medication and was terminated from the trial by the PI.
Irritability (Psychiatric disorders) | 2 (2) | 0 (0) — Subject discontinued medication and was terminated from the trial by the PI.
Study medication non compliance (Psychiatric disorders) | 3 (3) | 0 (0) — Subject discontinued medication and was terminated from the trial by the PI.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No